CLINICAL TRIAL: NCT00085332
Title: A Phase II Evaluation of Weekly Docetaxel (NSC #628503) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Docetaxel in Treating Patients With Recurrent or Persistent Endometrial Carcinoma (Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG-0129N; CDR0000368634
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well docetaxel works in treating patients with recurrent or persistent endometrial carcinoma (cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of docetaxel in patients with recurrent or persistent endometrial carcinoma.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 10-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrial carcinoma

  * Recurrent or persistent disease
  * Refractory to curative or standard therapy
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * At least 1 target lesion

    * Tumors within a previously irradiated field are not considered target lesions
* Received 1 prior chemotherapy regimen for endometrial carcinoma, including high-dose, consolidation, or extended therapy administered after surgical or non-surgical assessment

  * One additional non-cytotoxic regimen for recurrent or persistent disease allowed, including monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction
* Ineligible for a higher priority GOG protocol

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No neuropathy (sensory and motor) ≥ grade 2
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 3 weeks since prior biologic or immunologic therapy for malignant tumor
* No concurrent prophylactic growth factors
* No concurrent prophylactic thrombopoietic agents

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No more than 1 prior cytotoxic chemotherapy regimen (single or combination cytotoxic drugs)

Endocrine therapy

* At least 1 week since prior hormonal therapy for malignant tumor
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery

* Recovered from prior surgery

Other

* At least 3 weeks since other prior therapy for malignant tumor
* No prior anticancer therapy that would preclude current protocol therapy
* No concurrent amifostine or other protective reagents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Study Chair — Premiere Oncology
Locations (75):
- United States (71):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Women's Cancer Center - Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Cancer Center at Tufts - New England Medical Center, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - MD Anderson Cancer Center at University of Texas, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fletcher Allen Health Care - Medical Center Hospital of Vermont Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Australia New Zealand Gynaecological Oncology Trials Group, Camperdown, New South Wales, Australia
- Tom Baker Cancer Centre - Calgary, Calgary, Alberta, Canada
- Kagoshima City Hospital, Kagoshima, Japan
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Garcia AA, Blessing JA, Nolte S, Mannel RS; Gynecologic Oncology Group. A phase II evaluation of weekly docetaxel in the treatment of recurrent or persistent endometrial carcinoma: a study by the Gynecologic Oncology Group. Gynecol Oncol. 2008 Oct;111(1):22-6. doi: 10.1016/j.ygyno.2008.06.013. PMID 18675446